CLINICAL TRIAL: NCT03482336
Title: Munchy Monster: Using Video Gaming to Objectively Evaluate Front of Pack Labeling Strategies for School-aged Children
Brief Title: Using Video Gaming to Evaluate Front of Pack Labeling With Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura Bix, Professor, Michigan State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-678
Record Dates: First submitted 2017-09-18; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Child Obesity
Keywords: labeling; Front of pack; nutrition; nutrition facts panel
MeSH Terms: conditions — Pediatric Obesity | interventions — Color

STUDY DESIGN:
Intervention Model Description: Two blocks of participants were recruited. One block received no information regarding the FOP; for the second block, researchers pointed to an FOP and suggested that the information might be helpful in deciding which product was healthier.
Masking Description: Participants were handled differently in the methods. For the first block of participants, the FOP was not pointed out. For the second block, researchers merely pointed to the FOP and indicated that it might be helpful in decision making.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uninstructed Group (Other): For the first block of participants recruited (39, one of which withdrew from boredom), no overt reference was made regarding the FOP labels that were present on the images that participants viewed during the course of the video game. Participants comprising this block were referred to as "uninstructed."
  Interventions: Other: Four FOP label designs
- Minimally trained (Other): Realizing that subjects might not use the FOP during decision making when not informed that it contained nutrition information, we conducted a second experiment (N= 41) which provided minimal information about the FOP. These subjects (the "minimally instructed" group) were provided with further instruction. At the beginning of the experiment, in addition to being shown the basic premise of the game and told that Munchy preferred to eat healthy options, the researcher pointed to one of the FOPs and told children "this information might be helpful when you decide what's healthy."
  Interventions: Other: Four FOP label designs

INTERVENTIONS:
Other: Four FOP label designs — Color (present and absent) were crossed with facial icon (present and absent) for a total of four FOP label treatments. For each trial, both packages had the same FOP treatment, but one appeared at a "healthy level" while the second "unhealthy." Subjects were asked to choose the healthier option as quickly as possible. Accuracy and speed to correct selection both served as dependent variables.
  Other Names: color plus facial icon; no color plus facial icon; color plus no facial icon; no color plus no facial icon

SUMMARY:
Regulated nutrition information is complex, using decimal places and percentages. Front of pack (FOP) labels provide simplified nutrition information on the front of packages. It has been suggested that the traditional approach to nutrition labeling is difficult for children to use; this is unfortunate as childhood is a critical time for developing long-lasting eating habits and children influence purchase decisions.

Materials and Methods Children aged 6-10 played a video game in which participants fed "Munchy Monster" the healthier of two cereal products presented on a computer screen. Across trials the FOP format varied in a 2 (color/no color) x 2 (facial emotion icon/no facial icon) factorial design. Within a trial both cereals presented the same FOP format, with one cereal healthier than the other.

Results Data suggest that color coding and/or facial icon significantly benefits selection accuracy and speed, particularly for the youngest children. Minimal training (awareness of the FOPs existence and that it might contain nutrition information) further improved accuracy and speed of responses.

Conclusions FOPs that leverage visual indicators assist even young children in assessing the nutritional value of a product.

DETAILED DESCRIPTION:
Background It has been estimated that only two percent of children eat a diet that is consistent with the Food Guide pyramid, consuming diets that are too high in fat, saturated fat and sodium, and too low in fiber. Furthering concerns associated with these statistics is the fact that childhood is a determinant phase in the establishment of eating habits, and that developing healthy eating practices as a child has long-term health benefits.

That said, children are an attractive segment for food marketers. Children are not only represent a primary market with growing access to discretionary income, children also have significant power to influence decisions and are a promising future market. As such, kids represent an attractive target for marketers, and research suggests vulnerability to the messages which target them.

It has been suggested that directing messages to children "increases children's preferences for the foods advertised and increases their requests to parents for those foods." Recognizing this, packaging plays an important role in the marketing mix. The US Federal Trade Commission (FTC) has estimated that 12% of all youth marketing expenditures are spent on packaging and in-store in store display materials. This is because of packaging's ability to influence purchase within retail spaces, at the point where purchasing decisions are made; something researchers have referred to as the "nag factor."

Clearly, the idea of presenting information directed at children using packaging for the purpose of motivating sales is utilized; however, the idea of presenting regulated information (e.g. nutritional information) in a format that might be readily understood by this vulnerable audience has not been widely explored. A major goal of nutritional labeling on food packages is to help consumers make appropriate choices. However, the current approach to nutritional labeling is targeted at adults, rather than children.

Although children as young as age four are capable of classifying familiar foods (e.g. ice cream vs. broccoli) as healthy or unhealthy, the investigators are the first to examine whether children can use visual cues from Front of Pack (FOP) labels to compare and evaluate food products from the same category (cereal). FOP labels appear on the front of packages and provide truncated information about nutrients that tend to be associated with disease (e.g. fats, trans fats, sugar and sodium).

Two semi-directive overlays, namely, color (2 levels present/absent) and facial icon (present and absent) were crossed, for a total of four FOP treatments. The study investigated color because it represents the traffic light system, which is a standard FOP design in the United Kingdom (UK), and its use is a topic of significant debate globally. Investigators also tested the efficacy of schematic facial expressions representing relatively high, medium, and low values for nutrients (i.e. frowning for high; straight face for moderate and a smile for those low). Overwhelming evidence indicates that face stimuli are given extremely high attentional priority and that the processing of facial expressions of emotion requires very few cognitive resources. These findings suggest that a face stimulus might be a particularly effective stimulus for drawing attention to the FOP nutritional panel and conveying relative qualitative information about the nutritional value of a product. As such, study investigators postulated that FOP utilizing faces would be particularly well-suited for use with children. Faces are known for garnering increased attention in infants and children as young as age 4 can reliably identify facial expressions of emotion. In fact, developmental research often exploits children's ease of comprehending iconic faces to measure children's judgments of stimuli or situations.

Materials and Methods Investigators leverage these fundamental insights in work presented here, such insights can be used in ways that positively enhance attention to and understanding of nutrition information in a vulnerable audience, children aged 6 to 10.

Children were seated at a computer and given a brief overview of the game. The program began with an instruction scene in which a purple monster character (Munchy) said

"Hi my name is Munchy. I like to eat, but only healthy foods. Will you please feed me? In the game, you will see two cereal boxes. One is healthier than the other. To feed me please press the button on the side with the healthy cereal. If you select the healthy one I will eat it and you will get points. If you select the unhealthy one I will refuse to eat and you will not get any points. I am really hungry so please choose the healthy one as fast as you can. Do you have any questions?"

For each trial, both cereals had the same FOP treatment. However, one package contained "healthy levels" of key nutrients (e.g. for colored FOP three or more nutrients at "green levels") while the other contained "unhealthy levels" (three or more nutrients at "red levels"). Nutrients were categorized into high, moderate and low levels based on Traffic Light Label Guidelines released by the Food Standards Agency. The appearance of the brand and the position of the package (right or left side of screen) were randomized; additionally, a second randomization was done with the healthfulness level of the nutrition information such that the positioning (right side of screen or left) was randomized. As a result, for one subject brand X might appear as healthy, while for another it might be presented with unhealthy information. Each participant completed 80 trials, with each of the four FOP designs appearing in 20 trials per participant by the conclusion of the game. The time it took for the participant to make a correct choice was recorded along with a binary response of correct choice (yes or no).

Two blocks of participants were recruited. In the first block, no reference was made to the FOP labeling. For the second block of participants, at the beginning of the experiment, in addition to being shown the basic premise of the game and told that Munchy preferred to eat healthy options, the researcher pointed to one of the FOPs and told children "this information might be helpful when you decide what's healthy."

ELIGIBILITY:
Inclusion Criteria:

* 6-10 years of age
* Legally sighted
* have parent or legal guardian present (written consent of parent)
* have transportation to the test site
* be willing to share contact information for reminders be willing to have deidentified data stored provide written or verbal assent (depending on the age of the child)

Exclusion Criteria:

* legally blind
* no assent

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-04-12 (Actual)

PRIMARY OUTCOMES:
Proportion of Correct selections | During the one hour test period
  The correct selection of the healthier stimulus

SECONDARY OUTCOMES:
Time to correct selection | During the one hour test period
  The amount of time it takes to make a correct selection

CONTACTS AND LOCATIONS:
Overall Officials: Mark Becker, PhD, Principal Investigator — Michigan State University
Locations (1):
- School of Packaging, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
deidenitified file will be shared as supplemental file when published
Supporting Information: Analytic Code
Time Frame: Indefinitely upon publication
Access Criteria: will be shared as deidentified file upon publication